CLINICAL TRIAL: NCT03316716
Title: Peri-operative Active Warming Versus no Peri-operative Active Warming During Caesarean Section for Preventing Neonatal Hypothermia in Women Performing Skin-to-skin Care: A Randomized Controlled Trial
Brief Title: Active Warming Versus Non Active Warming During Caesarean Section for Preventing Neonatal Hypothermia
Acronym: NeoHyp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aliona Vilinsky-Redmond (Other)
Responsible Party: Sponsor-Investigator, Aliona Vilinsky-Redmond, Lead Investigator, The Rotunda Hospital
Organization: The Rotunda Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RotundaH
Record Dates: First submitted 2017-10-02; First posted 2017-10-20 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Neonatal Hypothermia
Keywords: caesarean section; neonatal hypothermia; maternal hypothermia; active warming; skin-to-skin contact

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Women randomised to the control group will receive the hospital's current standard of care which is the peri-operative administration of room-temperature (25°C) IV fluids (Hartman's solution) started before the insertion of regional anaesthesia and continued until the transfer of the woman to the postnatal ward.
- active warming group (Experimental): Women randomised in the intervention group will recieve warm IV fluids. The IV fluids (Hartman's solution) will be warmed to 39°C with the use of Hotline™ device.
  Interventions: Procedure: active warming

INTERVENTIONS:
Procedure: active warming — Women randomised to the intervention group will be administrated warm IV fluids (39°C) consisting of Hartman's solution with the use of the theatre's Hotline™ device. The Hotline™ device is set to 39°C in which the Hartman's solution bags will be infused to the women peri-operatively.
  Arms: active warming group

SUMMARY:
Peri-operative warming is well established for general operations, but there is limited literature on the active warming of pregnant women undergoing caesarean section (CS). Specifically, there is a lack of evidence on the effect, if any, of actively warming mothers on the new-born's temperature and general wellbeing. The two active warming methods recommended by NICE are the use of forced-air warming and fluid warmers.

Women's temperature tends to fall below the normal level (36.0oC to 37.5oC) during caesarean section if they have not been actively warmed during their operation (peri-operative). Peri-operative hypothermia may increase the morbidities experienced by women after caesarean section. While shivering is the most common postoperative incident, hypothermia may delay wound healing or increase the risk of wound infection, and can increase the risk of haemorrhage.

Neonatal hypothermia has a direct effect on the baby's cardiopulmonary, vascular system and central nervous system and increases the risks of mortality and morbidity. Specifically, neonatal hypothermia can lead to respiratory difficulties and apnoea, hypoxemia, carbon dioxide retention, metabolic acidosis, hypoglycaemia and decreased oxygen delivery to the tissues.

The absence of research and evidence on the effects of actively warming women undergoing caesarean section at term gestation on the temperature of new-borns during SSC means that further research is required.

DETAILED DESCRIPTION:
Peri-operative active warming is the practice of warming patients who undergo an operation with the use of one or more warming devices. Active warming can be initiated before, during and/or after an operation and its main purpose is to prevent and/or manage hypothermia in patients. Commonly used warming devices include: forced-air warming, fluid warmers, heating gel pads, water mattresses and electric blankets.

Peri-operative active warming has been researched over the past 30 years, with more sophisticated methods of active warming being introduced in recent years. Regardless of their complexity, these devices are used in order to prevent inadvertent perioperative hypothermia (IPH) and its complications in patients who undergo an operation. Complications of IPH include: thermal discomfort (including shivering), increased intra-operative blood loss, increased risk of wound infection, cardiac morbid events and increased length of stay in recovery room and in the hospital.

Although peri-operative warming is well established for general operations, there is a dearth of literature regarding active warming of pregnant women undergoing caesarean section (CS). The National Institute of Health and Care Excellence (NICE) developed guidelines for managing IPH for adults undertaking various general operations, however pregnant women and children/infants were excluded from these guidelines due to lack of evidence supporting or rejecting the use of peri-operative active warming for this population. The two active warming methods recommended by NICE include the use of forced-air warming and fluid warmers. Specifically all patients should be actively warmed with a forced-air warming device before/during their operation if their temperature is below 36°C and every patient should receive warmed IV fluids (via an IV fluid warmer) for volumes ≥500 mls of IV fluids. The patient's temperatures should be measured every 30 minutes from the time of their anaesthesia until their discharge to the ward.

An additional factor that complicates the decision of applying, or not, an active warming to pregnant women during a CS is the effect of active warming on new-borns during/after birth. This factor becomes even more relevant when skin-to-skin contact (SSC), between mothers and their new-borns, is initiated immediately after a CS. Specifically, there is a lack of research evidence on the effect, if any, of active warming on the new-born's temperature and general wellbeing. Three unpublished audits undertaken in the theatre department of a large maternity hospital in Dublin (between 2012 and 2014), have shown an increased number of hypothermic mothers and new-borns during and after CS. The hospital has a general practice of not actively warming pregnant women before/during their CS, and women at low risk for complications, usually perform SSC with their infants within minutes of birth. The more recent of these three audits (2014) showed that 86% (n=33) of women became hypothermic peri-operatively (defined as a core temperature below 36°C, while 35% (n=14) of the new-borns became mildly hypothermic after birth (defined as a core temperature below 36.5°C, after undergoing SSC, despite complying with the hospital guidelines.

SSC is a widely researched technique, in which a naked new-born (wearing only a nappy and a hat) is positioned on its mother's bare chest, covered with warm towels and a blanket. SSC has multiple advantages for both mothers and their new-borns. SSC is a usual practice within Rotunda Hospital, for babies born either vaginally or via CS. Although this technique is well established after vaginal birth, there is a great demand and attempts to establish it in mother-infant dyads after birth by a CS. A potential concern arising from this practice, however, is that new-borns, born by a CS, are more prone to losing their temperature and become hypothermic after a CS, compared with those born via normal birth. A risk factor is that if the mothers core temperature drops during the CS, leading to an even lower skin temperature, then the risk of a drop in the temperature of the new-born (via conduction) is increased by placing the naked baby for SSC on a mother whose temperature is suboptimal.

When either the mother or the new-born become hypothermic after a CS, there is a higher chance that both will be separated in order to be heated, often in different rooms. When this separation takes place, SSC is interrupted, early breastfeeding is delayed and the stress levels of the mother will increase as she would be concerned about her new-born's wellbeing. Additionally, babies who become hypothermic once, or have reoccurring cases of hypothermia, after birth are more likely to have invasive procedures such as blood sugar monitoring, rectal temperature measurements and blood checks for microbiological investigation and prophylactic administration of IV antibiotics (as per hospital's guidelines). These invasive procedures could be prevented especially in low risk babies (i.e. term babies with weight within the normal limits, or babies whose mothers are not diabetic) by keeping them warm and providing early feeding and SSC.

These obstacles could potentially be eliminated with the use of peri-operative active warming. The effects of peri-operative active warming in pregnant women remains inadequately researched, with even fewer studies evaluating the effects of peri-operative active warming on new-borns who are having SSC.

ELIGIBILITY:
Inclusion Criteria:

In order for women and their new-borns to be eligible to participate in the study they should be;

* Aged 18 years or over
* Able to provide informed consent for themselves and their babies
* Who have a singleton pregnancy between 37+0 and 41+6 weeks gestation
* Whose foetus/new-born is alive/born alive, and has no risk factors such as congenital or cardiovascular anomalies (see Appendix 2, TSRF)
* Who receive spinal or combined spinal anaesthesia for their caesarean section
* Have an elective CS
* Who are willing and able to perform skin-to-skin contact

Exclusion Criteria:

Women will be excluded from this study if they;

* Have pyrexia (> 37.5C on admission to ward)
* Have a maternal medical disease (ie. Spinal abnormalities, coagulation abnormalities, maternal serology positive, congestive heart failure, severe renal function impairment)
* Have general anaesthesia
* Have a baby who has a congenital anomaly (ie. Spina bifida, anencephaly, hydrocephaly, cardiovascular anomalies, anomalies of nervous system, defects of anterior abdominal wall)
* Have a baby who has abnormal Doppler artery velocimetry
* Have a stillbirth baby
* Have a recent USS estimating the fetal weight less than 2000g

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Neonatal hypothermia | approximately 50 minutes after delivery
  Neonatal hypothermia is defined as temperature < 36.5C

SECONDARY OUTCOMES:
Maternal Hypothermia | approximately 10 minutes before delivery
  Maternal hypothermia is defined as temperature < 36C
Maternal Hypothermia | approximately 30 minutes after delivery
  Maternal hypothermia is defined as temperature < 36C
Maternal Hypothermia | approximately 50 minutes after delivery
  Maternal hypothermia is defined as temperature < 36C
Maternal core temperatures | approximately 10 minutes before delivery
  Maternal core temperatures measured on 3 different occasions
Maternal core temperatures | approximately 30 minutes after delivery
  Maternal core temperatures measured on 3 different occasions
Maternal core temperatures | approximately 50 minutes after delivery
  Maternal core temperatures measured on 3 different occasions
Neonatal core temperatures | approximately 20 minutes after delivery
  Neonatal core temperatures measured on 2 different occasions
Neonatal core temperatures | approximately 50 minutes after delivery
  Neonatal core temperatures measured on 2 different occasions
Maternal thermal comfort | approximately 30 minutes after delivery
  Maternal thermal comfort measured using a 1-5 scale ranging from cold, cool, neutral, warm and hot
Shivering | approximately 30 minutes after delivery
  Shivering (yes/no)
additional maternal warming | approximately 30 minutes after delivery
  Use of additional warming of mothers (Bair Hugger™)
additional new-born warming | approximately 20 minutes after delivery
  Use of additional warming of new-born (incubator)
Occurrence of Adverse Events | From date of randomization until the date of first documented progression , assessed up to 2 hours post operation.
  Occurrence of Adverse Events during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Conan McCaul, MD, Principal Investigator — Head of Anaesthesia Department
Locations (1):
- Rotunda Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munday J, Hines S, Wallace K, Chang AM, Gibbons K, Yates P. A systematic review of the effectiveness of warming interventions for women undergoing cesarean section. Worldviews Evid Based Nurs. 2014 Dec;11(6):383-93. doi: 10.1111/wvn.12067. Epub 2014 Sep 30. PMID 25269994
- [Background] NICE (2008) The Management of Inadvertent Perioperative Hypothermia in Adults. Retrieved from http://www.ncbi.nlm.nih.gov/books/NBK53797/ on 18/8/2016.
- [Background] Vilinsky A., Sheridan A. & Nugent L.E. (2016) Preventing peri-operative maternal and neonatal hypothermia after skin-to-skin contact. Journal of Neonatal Nursing 22(4), 163-170.
- [Background] WHO (1997) Thermal protection of the newborn: a practical guide. , Maternal and Newborn Health/Safe Motherhood Unit, Division of Reproductive Health
- [Background] Knobel R, Holditch-Davis D. Thermoregulation and heat loss prevention after birth and during neonatal intensive-care unit stabilization of extremely low-birthweight infants. Adv Neonatal Care. 2010 Oct;10(5 Suppl):S7-14. doi: 10.1097/ANC.0b013e3181ef7de2. PMID 20838082
- [Background] Kumar V, Shearer JC, Kumar A, Darmstadt GL. Neonatal hypothermia in low resource settings: a review. J Perinatol. 2009 Jun;29(6):401-12. doi: 10.1038/jp.2008.233. Epub 2009 Jan 22. PMID 19158799
- [Background] Lunze K, Bloom DE, Jamison DT, Hamer DH. The global burden of neonatal hypothermia: systematic review of a major challenge for newborn survival. BMC Med. 2013 Jan 31;11:24. doi: 10.1186/1741-7015-11-24. PMID 23369256
- [Background] Smith J. (2014) Methods and Devices of Temperature Measurement in the Neonate: A Narrative Review and Practice Recommendations. Newborn and Infant Nursing Reviews 14(2), 64-71.
- [Background] Vilinsky A. & Sheridan A. (2014) Hypothermia in the newborn: An exploration of its cause, effect and prevention. British Journal of Midwifery 22(8), 557-562 556p.